CLINICAL TRIAL: NCT06818903
Title: Misoprostol Versus Intracervical Foley's Catheter for Termination of Second Trimester Abortion
Brief Title: Misoprostol in Missed Abortion
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ali Kamel Ali, Resident, Assiut University
Other Study IDs: A456743
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Abortion; Attempted
Keywords: Abortion; Misopristol; Foley catheter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Misopristol: women will be subjected to Foley catheter balloon insertion. A 16F Foley catheter will be inserted into the cervix and inflated with 40 ml of saline and it will be pulled out to ensure the balloon covered the internal os. The catheter will be fixed to the inner thigh with light traction .The Foley catheter balloon will be checked every 4 hours.
  Interventions: Drug: Misopristol
- Foley catheter: women will be subjected to Foley catheter balloon insertion. A 16F Foley catheter will be inserted into the cervix and inflated with 40 ml of saline and it will be pulled out to ensure the balloon covered the internal os. The catheter will be fixed to the inner thigh with light traction .The Foley catheter balloon will be checked every 4 hours. Women will be received, according to department policy,,At the same sitting 400μg misoprostol kept in posterior fornix and the dose will be repeated every three hours till the catheter got expelled out or till maximum five doses
  Interventions: Device: Foley catheter

INTERVENTIONS:
Drug: Misopristol — Foley catheter with Misopristol local application
  Other Names: Foley catheter
  Groups: Misopristol
Device: Foley catheter — Foley catheter alone
  Groups: Foley catheter

SUMMARY:
In this study we compare between the effectiveness of combined Foley's catheter with Misoprostol and intracervical Foley's catheter alone for termination of second trimester abortion.

DETAILED DESCRIPTION:
Termination of pregnancy (TOP) is defined as elective expulsion or extraction of products of conception from uterus instead of spontaneous onset of process irrespectable of duration of pregnancy. Worldwide mid-trimester abortion constitutes 10-15% of all induced abortions but responsible for two-thirds of all major complications Despite the recent advances in prenatal diagnosis in first trimester. Termination of pregnancy in second trimester due to foetal abnormalities and intrauterine foetal death still accounts for large number of abortions, and has increased the demand for rapid termination of pregnancy. In intrauterine fetal death in 2nd trimester, expulsion may take several weeks. This is associated with psychological trauma, coagulopathy and intrauterine infection. Among various methods of second trimester termination, evacuation and curettage induces risk of bleeding, infection, uterine perforation and cervical trauma. The introduction of misoprostol , a synthetic prostaglandin E1 analogue (PGE1) has become an important for cervical ripening and uterotonic action. It is economic, stable at room temperature and is associated with few side effects such as fever, vomiting and diarrhea. There is still debate about doses, routes and regimes of PGE1 for termination of pregnancy during 2nd trimester. It is active orally but more effective and better tolerated when administrated vaginally and has fewer side effects. Vaginal route is preferred in first and second trimester. The use of Foley's catheter has been recommended in many developing countries. The reports from different countries have mentioned excellent results with the use of Foley's catheter either alone or in combination with prostaglandins. The scope of our study: is to compare the use of Foley's catheter combination with Misoprostol versus Foley's catheter alone for pre induction cervical ripening and induction of second trimester abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 - 40 years of age with mid-trimester fetal death inutero.

  * Singleton pregnancies from 18-24 weeks.
  * women with unfavourable cervix (Bishop Score < 5) at the time of recruitment.
  * Previous one CS and non-previous CS pregnant women.

Exclusion Criteria:

* • Previous 2 CS or more.

  * Medical contraindications for prostaglandin therapy (allergy to prostaglandins or severe asthma).
  * co-morbidities like severe anemia (Hb < 7g/dl), hypertension, diabetes, or coagulopathy .
  * Women with excessive vaginal discharge or rupture of membrane.
  * Women having any complication in previous caesarean like endometritis, reopening, scar dehiscence etc.
  * Active genital infection e. g. active genital Herpes simplex infection.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women who are indicated for termination of pregnancy in second trimester due to fetal abnormalities and intrauterine fetal death
Sampling Method: Non-Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Interval time | periprocedurally
  the interval (hours) between Foley catheter balloon insertion to complete abortion

IPD SHARING:
Plan to Share IPD: Undecided